CLINICAL TRIAL: NCT00725569
Title: Effect of Homeopathic Drugs Bellis Perennis ו- Staphysagria on the Post-operative Recovery, of Women Undergoing Cesarean Section- (an Exploratory) Double Blind, Placebo Controlled Study
Brief Title: Homeopathy for Post-operative (C. Section) Recovery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Menachem Oberbaum, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POR2008
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Cesarean Section
Keywords: Caesarian Section; Homeopathy; Pain; Analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Bellis perennis and Staphysagria (C6)
  Interventions: Drug: Bellis perennis and Staphysagria (C6)
- B (Active Comparator): Bellis perennis and Staphysagria (C30)
  Interventions: Drug: Bellis perennis and Staphysagria (C30)
- C (Placebo Comparator): Placebo Remedy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bellis perennis and Staphysagria (C6) — homeopathic remedy
  Arms: A
Drug: Bellis perennis and Staphysagria (C30) — Homeopathic Remedy
  Arms: B
Drug: Placebo — Placebo remedy, identical in size, shape and taste to treatment remedies
  Arms: C

SUMMARY:
The planned study will be conducted in a prospective, randomized, double blind placebo controlled manner. Two "anti-traumatic" Homeopathic remedies (Arnica montana and Staphysagria) will be used. The selection of these remedies was based on a previous trial that showed a statistical difference in Hemoglobin levels favoring pregnant women treated with these drugs following delivery.

The proposed study will focus on the post-operative recovery of women undergoing Cesarean section. According to Homeopathic principles, these two remedies are believed to improve the "vital force", and will therefore improve convalescence following surgery in the study group. The study will include 90 women between the ages of 18 and 50 years who are scheduled for elective Cesarean Section. Exclusion criteria are: obesity (above 100kg), malignancy, psychiatric illness, diabetes and multipara pregnancies. Participants will be inducted following a detailed explanation by an MD and signing of an informed consent form, and then subdivided randomly into three groups numbering 30 in each: Two groups will be treated with homeopathic drugs of varied doses, and the third will get a placebo remedy which is indistinguishable from the other drugs. Outcome measures will include: 1. Blood loss - as estimated by a reduction in serum Hemoglobin levels. 2. Pain -to be evaluated by a numerical rating score (NRS) 3. Analgesic use 4. Length of post-operative stay and complications. 5. Quality of life outcomes - to be assessed using the MOS SF-36 questionnaire at one and four weeks following surgery. Although not expected, adverse events will be monitored.

If, as we anticipate, the homeopathic treatment proves to be both safe and effective in shortening the duration of post-operative healing, this will have significant implications, with respect to both healthcare costs and patient suffering. It will also open the door for further research in the field of trauma medicine, as well as other stress-related illness.

ELIGIBILITY:
Inclusion Criteria:

* women hospitalized for elective C. Section, from the 1st to 3rd pregnancies.
* Age < 50 years
* Body weight < 100 kg
* Signing of informed consent form

Exclusion Criteria:

1. suspected/proven malignancy
2. underlying Axis-1 psychiatric illness
3. age < 18 years
4. diabetes mellitus (NIDDM/IDDM)
5. unable to comply with study proceedings

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
pain, to be evaluated using a numerical rating score (NRS) on a 100mm scale (0= no pain whatsoever, 100 = unbearable pain). | 4 weeks

SECONDARY OUTCOMES:
Analgesic Use | 4 weeks
Duration of Hospital Stay | 4 weeks
Time from Surgery to First Bowel Movement | 4 days
Blood Loss | 4 days
Post-operative Complications the following complications will be noted: Nausea, vomiting, abdominal distension, fever, urinary tract infection, thrombophlebitis, wound infection, wound hematoma, ileus, vaginal bleeding. | 4 weeks
Quality of Life Assessment | 4 weeks
Adverse Effects of Treatment | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021